CLINICAL TRIAL: NCT04407988
Title: Phase II Study of Pyrotinib in Combination With Letrozole in Patients With HER2-Positive, ER-Positive Metastatic Breast Cancer
Brief Title: Pyrotinib in Combination With Letrozole in Patients With HER2-Positive, ER-Positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-008
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: Pyrotinib plus Letrozole
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib plus Letrozole (Experimental)
  Interventions: Drug: Pyrotinib Maleate plus Letrozole

INTERVENTIONS:
Drug: Pyrotinib Maleate plus Letrozole — pyrotinib(400 mg once daily) + Letrozole (2.5 mg once daily)

SUMMARY:
This is a prospective, single-arm, multi-center clinical study of pyrotinib in combination With letrozole in patients With HER2-Positive, ER-Positive metastatic breast cancer. Our aim was to explore the efficacy and safety of pyrotinib combined with letrozole in patients with HER2-positive, ER-positive metastatic breast cancer.

DETAILED DESCRIPTION:
ER+/HER2+ metastatic breast cancer is a special subtype of HER2+ breast cancer. General guidelines recommend chemotherapy combined with HER2-targeted therapy for this subtype of patients. However, for the highly selected patients with ER- positive/HER2-positive ABC, ET + anti-HER2 therapy could be chosen as first-line therapy. And Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. Therefore this study is planned to enroll 86 patients with HER2-positive, ER-positive metastatic breast cancer receiving first-line treatment with pyrotinib and letrozole. The main purpose was to evaluate the efficacy and safety of pyrotinib combined with letrozole in patients with HER2-positive, ER-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HER2+/ER+ recurrent or metastatic breast cancer confirmed by histopathology;

   * HER2 positive: HER2 IHC 3+, or HER2 IHC 2+ and ISH positive
   * ER positive: the percentage of cells positive for ER expression ≥ 10%
2. Premenopausal, perimenopausal or postmenopausal patients (with OFS, if pre- or perimenopausal);
3. If the patient is bilateral breast cancer, metastasis lesions must be HER2 and ER positive;
4. 18-70 years old;
5. ECOG PS 0～1;
6. Life expectancy is not less than 12 weeks;
7. At least one measurable lesion according to RECIST 1.1;
8. Prior (neo) adjuvant trastuzumab, pertuzumab or chemotherapy were eligible, and the disease free interval must be greater than 12 months from completion of (neo) adjuvant trastuzumab and pertuzumab to metastatic diagnosis;
9. Prior (neo) adjuvant hormone therapy was allowed, if received adjuvant AI, the disease free interval must be greater than 12 months from the completion of treatment;
10. Disease-free Survival after surgery (DFS) ≥12 months;
11. Patients with adequate organ function before enrollment: ANC ≥ 1.5×109/L, PLT ≥ 75×109/L, Hb ≥ 100 g/L; TBIL≤1.0ULN；ALT and AST≤3×ULN (ALT and AST≤5×ULN if liver metastasis); BUN and Cr≤1.5×ULN and CCr≥50 mL/min; LVEF ≥ 50% and QTc < 480 ms;
12. Signed informed consent.

Exclusion Criteria:

1. Central nervous system metastasis;
2. patients with Visceral crisis;
3. Unable to swallow, chronic diarrhea and intestinal obstruction, there are many factors affecting drug use and absorption;
4. received radiotherapy, hormone therapy, chemotherapy, surgery (excluding local puncture) or molecular targeted therapy for advanced or metastatic disease;
5. received radiotherapy, chemotherapy, surgery (excluding local puncture) or molecular targeted therapy within 4 weeks prior to randomization;
6. Received hormone therapy within 2 weeks prior to randomization;
7. Participated in other clinical trial within 4 weeks prior to randomization;
8. Previous or ongoing use of HER2-targeted tyrosine kinase inhibitors (lapatinib, neratinib or pyrotinib);
9. Other malignancies within 5 years, except for cured skin basal cell carcinoma,carcinoma in-situ of uterine cervix and squamous-cell carcinoma;
10. Receive other anti-tumour therapy at the same time;
11. History of immunodeficiency, including HIV positive, HCV, active hepatitis B, or other acquired, congenital immunodeficiency disorders, or organ transplantation, is known;
12. History of any kind of Heart disease;
13. All female patients in pregnancy or breastfeeding period, fertile women with positive baseline pregnancy tests;
14. Evidence of significant medical illness that will substantially increase the risk on the participation or completion of the study in the investigator's judgment. Examples included, but not limited to, hypertension, severe diabetes, etc;
15. History of neurological or psychiatric disorders, including epilepsy or dementia;
16. Patients not eligible for this study judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit rate (CBR) | Estimated 12 months
  Ratio of CR,PR and SD greater than or equal to 24 weeks in all subjects

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Estimated 12 months
  Ratio of CR and PR in all subjects
Progression Free Survival (PFS) | Estimated 12 months
  From enrollment to progression or death (for any reason
Overall Survival (OS) | Estimated 24 months
  From enrollment to death (for any reason)
Adverse Events and Serious Adverse Events | From informed consent through 28 days following treatment completion
  Adverse events are described in terms of CTC AE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Quchang Ouyang, PhD, Principal Investigator — Department of Breast Cancer Medical Oncology
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Hu ZY, Yan M, Xiong H, Ran L, Zhong J, Luo T, Sun T, Xie N, Liu L, Yang X, Xiao H, Li J, Liu B, Ouyang Q. Pyrotinib in combination with letrozole for hormone receptor-positive, human epidermal growth factor receptor 2-positive metastatic breast cancer (PLEHERM): a multicenter, single-arm, phase II trial. BMC Med. 2023 Jun 26;21(1):226. doi: 10.1186/s12916-023-02943-2. PMID 37365596